CLINICAL TRIAL: NCT02966132
Title: Interactive Mobile Doctor (iMD) for Asian Smokers
Acronym: iMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Asian Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRDRP 24AT-1301; 24AT-1300 (Other Grant/Funding Number: TRDRP)
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Smoking Cessation
Keywords: Asian American; Immigrant Health; Digital Health Intervention; Federally Qualified Health Centers
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- iMD (Experimental): Participants will receive interactive "Mobile Doctor" (iMD) intervention in English, Chinese, Korean or Vietnamese languages that delivers video education tailored to patient's responses on a computer tablet during the clinic visit to enhance patient-provider discussion of tobacco use. The iMD intervention implements the 5As (Ask, Advice, Assess, Assist, and Arrange) recommended by the Clinical Practice Guideline for treating tobacco dependence. A summary printout including provider recommendation options, brief summary of smoking status, quit intention and concerns are provided to patients to empower them to discuss tobacco use with their providers.
  Interventions: Behavioral: iMD
- NPA (Active Comparator): Participants will receive a video education providing nutrition and physical activity recommendations right before before seeing their providers. A printout summarizing topics presented in the education videos will be provided to the patient
  Interventions: Behavioral: NPA

INTERVENTIONS:
Behavioral: iMD — Interactive video education delivered on a tablet computer
  Arms: iMD
Behavioral: NPA
  Arms: NPA

SUMMARY:
The primary aim of the proposed study is to conduct a randomized controlled trial (RCT) to evaluate the efficacy of the Interactive Mobile Doctor (iMD) intervention targeting 150 Chinese-, Korean- or Vietnamese-speaking male patients who smoke daily and have a scheduled clinic visit at Asian Health Services primary care.

DETAILED DESCRIPTION:
The Asian American population is the fast-growing racial group during 2000 and 2010. Smoking prevalence among that Vietnamese (43%), Chinese (32%), and Korean (27%) men who spoke limited English are disproportionately higher than that of men of all races combined (17%). Thus, some Asian groups, including Chinese, Korean and Vietnamese, have an unequal burden of tobacco-related diseases. Asian Health Services (AHS) is a federally-qualified health center in Alameda County, California, providing services in English and 12 different Asian languages. The vast majority of the patients are Chinese, Vietnamese, and Korean with low income. Because of high smoking rates and associated health impacts on patients and their families, promoting smoking cessation is a health priority for AHS. The Vietnamese Community Health Promotion Project (VCHPP) at UCSF has conducted numerous intervention studies to promote smoking cessation among Asian Americans. Given the shared research interest, AHS and VCHPP have partnered to address smoking in Asian Americans. The partners received a TRDRP pilot Community-Academic Research Award grant to develop an interactive "Mobile Doctor" (iMD) intervention in Korean and Vietnamese languages that delivers video education tailored to patient's responses on a computer tablet during the clinic visit to enhance patient-provider discussion of tobacco use. The primary goal of the proposed study is to evaluate the iMD intervention with an expansion to the Chinese language in its efficacy to promote patient-provider discussion and quitting smoking in Chinese, Korean, and Vietnamese male smokers. The study will enroll 150 AHS Chinese-, Korean- or Vietnamese-speaking patients who smoke daily and have a scheduled clinic visit. Participants will then be assigned (by chance) into either receiving 1) iMD on tobacco or 2) video education on nutrition and physical activity recommendations. Participants will be assessed at: before the scheduled intervention visit, immediately after or within one week of the intervention visit, and 6 months following the intervention visit. Additional data will be obtained from EHR. The investigators anticipate that, when compared to participants receiving usual care alone, those who receive the iMD will be more likely to receive physician advice on their tobacco use both at their intervention visit and at one visit following the intervention visit within 6 months as documented in EHR; and at 6 months follow-up, those receiving the iMD will be more likely to report having been able to quit smoking for at least one day during the study period, and to have reported having quit smoking for at least 7 days with their abstinence status verified using a saliva sample. The long-term goal is to understand effective ways to enhance patient-provider communication in tobacco use and to leverage each clinic encounter in promoting smoking cessation among patients in community health settings.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older;
* male;
* English, Chinese- (Cantonese), Korean- or Vietnamese-speaking;
* self-identified as ethnic Chinese, Korean, Vietnamese or Asian
* current smoker as identified by EHR;
* have an already scheduled provider visit at Asian Health Services;
* smoke at least 1 cigarette daily in the last 7 days; and
* unwilling or unavailable to participate the in study procedures (e.g., to complete a brief post-visit survey right after the visit or by phone) according to the group assignment

Exclusion Criteria:

* Have vision and/or hearing difficulty that prevents the participant from viewing or hearing the intervention video messages and/or completing the assessment in person or by telephone

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
abstinence | 6-month
  7-day point prevalent smoking abstinence biochemically verified by salivary cotinine
quite attempt | 6-month
  self-reported 24-hour quit attempts

SECONDARY OUTCOMES:
patient-provider discussion | immediate post-intervention
  self-reported by patient whether discussion on tobacco use took place at the intervention clinical encounter
EHR documented 5As | immediate post-intervention
  EHR progress notes documenting delivery of the clinical guideline

CONTACTS AND LOCATIONS:
Overall Officials: Thu Quach, PhD, Principal Investigator — Asian Health Services; Janice Tsoh, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Asian Health Services, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data available at this time.

REFERENCES:
- [Derived] Tsoh JY, Quach T, Duong TB, Sa Nan Park E, Wong C, Huang SM, Nguyen TT. Interactive Mobile Doctor (iMD) to Promote Patient-Provider Discussion on Tobacco Use among Asian American Patients in Primary Care: A Pilot Study. J Am Board Fam Med. 2018 Nov-Dec;31(6):869-880. doi: 10.3122/jabfm.2018.06.180018. PMID 30413543